CLINICAL TRIAL: NCT07255846
Title: A Phase 1 Trial of TER-1754 in Patients With Hereditary Hemorrhagic Telangiectasia
Brief Title: A Trial of TER-1754 in Patients With Hereditary Hemorrhagic Telangiectasia
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Terremoto Biosciences Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TER-1754-C01
Record Dates: First submitted 2025-11-14; First posted 2025-12-01 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Hereditary Hemorrhagic Telangiectasia (HHT)
Keywords: Hereditary hemorrhagic telangiectasia; ENG, ACVRL1/ALK-1 alterations; Osler-Weber-Rendu; HHT; Anemia; Nosebleed; Epistaxis; AVM; Arteriovenous Malformation
MeSH Terms: conditions — Telangiectasia, Hereditary Hemorrhagic; Anemia; Epistaxis; Arteriovenous Malformations

STUDY DESIGN:
Intervention Model Description: Phase 1a is an open-label dose-escalation trial. Phase 1b is a 3-arm randomized placebo-controlled design. The Phase 1b treatment period is separated into a blinded treatment segment followed by an open-label extension (OLE) segment
Masking Description: Phase 1a is open label, dose escalation. The Phase 1b treatment period is separated into a blinded treatment segment followed by an open-label extension (OLE) segment
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Phase 1a (Dose Escalation) TER-1754 dose escalation (Experimental): TER-1754 Oral tablets
  Interventions: Drug: TER-1754
- Phase 1b (Proof of Concept) (Placebo Comparator): Placebo oral tablets
  Interventions: Drug: Placebo
- Phase 1b (Proof of Concept) - Phase 1b TER-1754 lower dose to begin post determination in Phase 1a (Experimental): Patient will receive one of the two doses determined post Phase 1a
  Interventions: Drug: TER-1754
- Phase 1b (Proof of Concept) - Phase 1b TER-1754 higher dose to begin post determination in Phase 1a. (Experimental): Patient will receive one of the two doses determined post Phase 1a
  Interventions: Drug: TER-1754

INTERVENTIONS:
Drug: TER-1754 — QD or BID, orally in 28-day cycles
  Arms: Phase 1a (Dose Escalation) TER-1754 dose escalation
Drug: Placebo — Number of tablets will be confirmed post Phase 1a
  Arms: Phase 1b (Proof of Concept)
Drug: TER-1754 — Phase 1b dose to be determined post Phase 1a
  Arms: Phase 1b (Proof of Concept) - Phase 1b TER-1754 higher dose to begin post determination in Phase 1a.; Phase 1b (Proof of Concept) - Phase 1b TER-1754 lower dose to begin post determination in Phase 1a

SUMMARY:
This is a Phase 1a/1b, multicenter study evaluating the safety, tolerability, pharmacokinetics, pharmacodynamics, and clinical activity of TER-1754 (a novel AKT1 inhibitor) in patients with HHT.

DETAILED DESCRIPTION:
This is a first-in-human, Phase 1, multicenter trial that includes two parts:

* Phase 1a (dose escalation) will evaluate the safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD), and preliminary clinical activity of TER-1754 in patients with HHT and determine the maximum tolerated or administered dose.
* Phase 1b (proof of concept) will evaluate clinical activity and further characterize the safety profile of TER-1754 in patients with HHT. The Phase 1b treatment period is separated into a blinded treatment segment followed by an open-label extension (OLE) segment.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide a signed and dated written informed consent prior to any study-specific procedures, sampling, or data collection.
* A clinical diagnosis of HHT as defined by the Curaçao criteria
* Baseline (1-month) ESS ≥ 4
* ECOG ≤ 2
* Anemia or parental iron infusion of at least 500 mg or transfusion of at least 2 units of RBCs within the preceding 24 weeks.
* Adequate bone marrow function
* Adequate renal function
* Adequate hepatic function

Exclusion Criteria:

* Prior nonresponse or loss of response to an agent that inhibits AKT1 and/or AKT2 as the primary mechanism of action.
* Diagnosis of DM requiring insulin treatment
* Known significant bleeding sources other than nasal, GI, or menstrual/ uterine
* Known underlying hypoproliferative anemia or clinically significant hemolytic anemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-12-15 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Phase 1a: Safety and Tolerability of TER-1754 | up to 48 weeks
  Incidence of adverse events characterized by type, seriousness, relationship to study treatment, and severity according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE) v5.0
Phase 1a: Maximum Tolerated Dose (MTD) and/or Maximum Administrated Dose (MAD) of TER-1754 | 28 days
  Incidence dose-limiting toxicities (DLTs) characterized by type, seriousness, and severity according to NCI CTCAE v5.0 (dose escalation only).
Phase 1b - Evaluate the Change from baseline in epistaxis and symptom-related clinical activity scores at Week 24 | 48 weeks
  Assess change from baseline in epistaxis duration

SECONDARY OUTCOMES:
Phase 1a and 1b: Evaluate TER-1754 Peak Plasma Concentration (Cmax) | up to 48 weeks
  Cmax of TER-1754 following single and multiple dosing.
Phase 1a and 1b: Evaluate change from baseline in Daily Epistaxis (EQ) Questionnaire | up to 48 weeks
  Change from baseline in EQ Questionnaire based on patient self-reported epistaxis frequency, severity and duration, where:
  Epistaxis frequency: number of epistaxis events per week Epistaxis duration: total minutes of bleeding Epistaxis intensity - From mild to severe: Spotting, dripping, dripping quickly, steady stream, pouring, and gushing.
Phase 1a and 1b: Evaluate HHT-specfic quality of life | Up to 48 weeks
  Change from baseline in HHT-specific QoL (HHT-QoL), where The total score ranges from 0 (no limitations) to 16 (severe limitations).
Phase 1a and 1b: Evaluate TER-1754 Time to Peak Concentration (Tmax) | Up to 48 weeks
  Time at which maximum observed plasma concentration occurs.
Phase 1a and 1b: Evaluate TER-1754 Area Under the Concentration-Time Curve (AUC0-last) | Up to 48 weeks
  Area under the plasma concentration-time curve from time zero to last measurable concentration (AUC0-last)
Phase 1a and 1b: Evaluate TER-1754 AUC0-24 | Up to 48 weeks
  Area under the plasma concentration-time curve from time zero to 24 hours (AUC0-24)
Phase 1a and 1b: Evaluate TER-1754 AUC∞ | Up to 48 weeks
  Area under the plasma concentration versus time curve extrapolated to infinity (AUC∞) of TER-1754 following single and multiple dosing.
Phase 1a and 1b: Evaluate TER-1754 Terminal Half-Life (t½) | Up to 48 weeks
  Terminal elimination half-life (t½) of TER-1754 calculated from the terminal slope of the plasma concentration versus time profile.
Phase 1a and 1b: Evaluate TER-1754 Mean Residence Time (MRT) | Up to 48 weeks
  Mean residence time (MRT) of TER-1754.
Phase 1a and 1b: Evaluate TER-1754 Accumulation Ratio at Steady State | Up to 48 weeks
  Accumulation ratio of TER-1754 at steady state, calculated as the ratio of exposure at steady state to exposure after the first dose.
Phase 1a and 1b: Change from baseline in Nasal Obstruction Symptom Evaluation Score for HHT (NOSE HHT) | up to 48 weeks
  Change from baseline in the NOSE HHT score, a validated scale measuring nasal obstruction in HHT. The score ranges from 0 to 4, with higher scores indicating more severe symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Innovative Hematology, Inc., Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No